CLINICAL TRIAL: NCT07163624
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group Phase II Study to Evaluate the Efficacy and Safety of UBT251 Injection in Patients With Type 2 Diabetes Mellitus
Brief Title: UBT251 Injection Phase II (Type 2 Diabetes Mellitus) Study
Acronym: T2DM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The United Bio-Technology (Hengqin) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUL-UBT251(Ⅱ-2)202405; CTR20250029 (Other: National Medical Products Administration)
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- UBT251 Injection 2.0 mg (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 0.5 mg subcutaneous injection with increasing doses at 5, 9weeks to 1.0 mg and 2.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 2.0 mg and UBT251 Injection Placebo
- UBT251 Injection 4.0 mg（ID 0.5 mg） (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 0.5 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 1.0 mg, 2.0 mg and 4.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 4.0 mg (ID 0.5 mg) and UBT251 Injection Placebo
- UBT251 Injection 4.0 mg（ID 1.0 mg） (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 1.0 mg subcutaneous injection with increasing doses at 5 and 9 weeks to 2.0 mg and 4.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 4.0 mg (ID 1.0 mg) and UBT251 Injection Placebo
- UBT251 Injection 6.0 mg (Experimental): Each subject will receive UBT251 Injection and UBT251 Injection Placebo, s.c. once weekly for 24 weeks. The starting dose of UBT251 Injection will be 1.0 mg subcutaneous injection with increasing doses at 5, 9 and 13 weeks to 2.0 mg, 4.0 mg and 6.0 mg once weekly.
  Interventions: Drug: UBT251 Injection 6.0 mg and UBT251 Injection Placebo
- Semaglutide Injection （Ozempic®）1.0 mg (Active Comparator): Each subject will receive Semaglutide Injection （Ozempic®）, s.c. once weekly for 24 weeks. The starting dose of Semaglutide Injection （Ozempic®） will be 0.25 mg subcutaneous injection with increasing doses at 5 and 9 weeks to 0.5 mg and 1.0 mg once weekly.
  Interventions: Drug: Semaglutide Injection (Ozempic®)

INTERVENTIONS:
Drug: UBT251 Injection 2.0 mg and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo once weekly
  Arms: UBT251 Injection 2.0 mg
Drug: UBT251 Injection 4.0 mg (ID 0.5 mg) and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo once weekly
  Arms: UBT251 Injection 4.0 mg（ID 0.5 mg）
Drug: UBT251 Injection 4.0 mg (ID 1.0 mg) and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo once weekly
  Arms: UBT251 Injection 4.0 mg（ID 1.0 mg）
Drug: UBT251 Injection 6.0 mg and UBT251 Injection Placebo — UBT251 Injection and UBT251 Injection Placebo once weekly
  Arms: UBT251 Injection 6.0 mg
Drug: Semaglutide Injection (Ozempic®) — Semaglutide Injection (Ozempic®) once weekly
  Arms: Semaglutide Injection （Ozempic®）1.0 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy of UBT251 injection after 24 weeks of continuous administration in patients with type 2 diabetes mellitus and to recommend the dosing regimen for the Phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years (inclusive) at the time of informed consent; sex not restricted.
* Documented diagnosis of type 2 diabetes mellitus with HbA1c ≥7.0% and ≤10.5% at screening.
* Lifestyle intervention or stable-dose metformin treatment (≥1000 mg/day) for at least 3 months before screening; "stable" defined as no change in daily dose during this period.
* Body weight: ≥50.0 kg for men and ≥45.0 kg for women at screening; body-mass index (BMI) 23.0-40.0 kg/m² (inclusive).
* Subject (and partner) agrees to use effective contraception from screening until 6 months after study completion and has no plans to donate sperm or ova during this period.
* Has been fully informed about the study and voluntarily signed the written informed consent form.

Exclusion Criteria:

* Known hypersensitivity to the investigational product or any of its excipients, to other GLP-1 receptor agonists, or history of clinically significant multiple or severe drug allergies; current allergic disease, high allergic disposition, or history of anaphylaxis.
* Prior use of any of the following medications:

  1. Any antihyperglycemic agent other than metformin within 3 months before screening, including GLP-1 analogues, oral antidiabetics, insulin, Chinese herbal medicines or health products with glucose-lowering effects.
  2. Systemic glucocorticoids, growth hormone, or any drug that may affect glucose metabolism within 3 months before screening.
  3. Any weight-loss medication within 3 months before screening.
* History or evidence of any of the following conditions:

  1. Diabetes other than type 2 (e.g., type 1 diabetes, specific types of diabetes).
  2. Acute or chronic pancreatitis, or history of pancreatic surgery.
  3. Symptomatic gallbladder disease within 2 years before screening (imaging-confirmed gallstones with physician-diagnosed related abdominal pain); subjects with prior cholecystectomy without sequelae may be included.
  4. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
  5. Hematologic disorders that may interfere with HbA1c measurement or increase subject risk, or any disease causing hemolysis or red-cell instability.
  6. History of depression or severe psychiatric disorders including suicidal ideation/attempt, schizophrenia, or bipolar disorder.
  7. Clinically significant active cardiovascular or cerebrovascular disease within 6 months before screening: myocardial infarction or unstable angina; cardiac surgery; congestive heart failure; cerebrovascular accident including stroke/TIA; any other cardiovascular/cerebrovascular condition deemed unsuitable by the investigator.
  8. Retinopathy requiring urgent treatment at screening.
  9. History of severe hypoglycemic coma or recurrent hypoglycemia within 2 months before randomization.
  10. Diabetic acute metabolic complications or diabetic foot within 6 months before screening.
  11. Gastroparesis or other disorders associated with delayed gastric emptying, uncontrolled gastro-esophageal reflux disease, or any gastrointestinal condition that, in the investigator's opinion, increases risk after study drug administration.
  12. Major surgery, severe trauma, or severe infection within 1 month before screening judged by the investigator to preclude study participation.
  13. History of malignancy (except adequately treated basal-cell carcinoma or carcinoma in situ of the cervix).
  14. Concurrent medical conditions (neurologic, endocrine, psychiatric, etc.) that, in the investigator's opinion, could compromise subject safety, affect efficacy assessments, or interfere with compliance.
* Clinically significant abnormal findings at screening, including:

  1. Fasting C-peptide <0.81 ng/mL.
  2. Hepatic or renal impairment: ALT and/or AST ≥2.5×ULN; total bilirubin ≥1.5×ULN; eGFR <60 mL·min-¹·1.73 m-².
  3. Serum calcitonin ≥50 pg/mL.
  4. Unstable thyroid medication requirement or clinically significant abnormal thyroid function tests necessitating new treatment.
  5. Fasting triglycerides ≥5.6 mmol/L.
  6. Serum amylase and/or lipase >2.0×ULN.
  7. INR above the upper limit of normal.
  8. Hemoglobin <110 g/L (males) or <100 g/L (females).
  9. Uncontrolled or untreated hypertension.
  10. Clinically significant ECG abnormalities: second- or third-degree AV block; long-QT syndrome or QTcF >470 ms (female) or >450 ms (male); pre-excitation syndrome; or any severe arrhythmia requiring treatment.
  11. Any physical examination, vital sign, or laboratory abnormality that, in the investigator's judgment, poses significant risk to the subject or may interfere with safety, PK, or PD evaluations.
* Positive tests for:

  * HBsAg with HBV DNA above the reference range;
  * Anti-HCV with HCV RNA above the ULN;
  * HIV antibody;
  * Treponemal antibody (syphilis).
* Blood loss or donation >400 mL, or receipt of blood/blood products within 3 months before screening; hemoglobinopathy, hemolytic anemia, or sickle-cell disease.
* Participation in another clinical trial within 3 months before screening.
* History of alcohol or drug abuse; alcohol abuse defined as >14 standard drinks per week (men) or >7 (women).
* Pregnant or lactating women.
* Inability to tolerate venipuncture, or history of vasovagal syncope or severe needle phobia.
* Any other condition that, in the investigator's opinion, renders the subject unsuitable for the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2025-03-22 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c at Week 24 | Baseline to week 24
  HbA1c was obtained at baseline and at Week 24

SECONDARY OUTCOMES:
Change Change from baseline to week 12, 16, 20 in HbA1c | Week 12, 16, 20
  HbA1c was obtained at baseline and at Week 12, 16, 20
Change in venous fasting plasma glucose (FPG) from baseline to week 12, 16, 20, 24 | Week 12, 16, 20, 24
  FPG was obtained at baseline and at Week 12, 16, 20, 24
Change in 2-hour post-standard-meal plasma glucose from baseline to week 12, 24 | Week 12, 24
  2-hour post-standard-meal plasma glucose was obtained at baseline and at Week 12, 24
Change in body weight from baseline to week 12, 24 | Week 12, 24
  Body Weight was obtained at baseline and at Week 12, 24
Change in waist circumference from baseline to week 12, 24 | Week 12, 24
  Waist circumference was obtained at baseline and at Week 12, 24
HbA1c target achievement rates (<7.0%) at Week 24 | Week 24
  Percentage of participants who achieved HbA1c <7.0% is presented
HbA1c target achievement rates (≤6.5%) at Week 24 | Week 24
  Percentage of participants who achieved HbA1c ≤6.5% is presented
FPG target achievement rate (4.4-7.0 mmol/L) at Week 24 | Week 24
  Percentage of FPG target achievement (4.4-7.0 mmol/L) at Week 24
Combined target achievement rate for both HbA1c and FPG at Week 24 | Week 24
  Percentage of Combined target achievement rate for both HbA1c and FPG at Week 24
Change from baseline to week 24 in fasting lipid profile | Week 24
  Fasting lipid profile was obtained at baseline and at Week 24
Change from baseline to week 24 in systolic blood pressure | Week 24
  Systolic blood pressure was obtained at baseline and at Week 24
Change from baseline to week 24 in diastolic blood pressure | Week 24
  Diastolic blood pressure was obtained at baseline and at Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- The United Bio-Technology (Hengqin) Co., Ltd., Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No